CLINICAL TRIAL: NCT07041086
Title: Prehospital ECPR in Moravia Silesia Region - Assessing the Effectiveness, Feasibility and Time of ECPR by Simulating Connections and Real Interventions.
Brief Title: Prehospital ECPR in Moravia Silesia Region
Acronym: 01-Pain
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: Emergency Medical Services, Moravian-Silesian Region (Unknown)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-01-Pain
Record Dates: First submitted 2025-06-12; First posted 2025-06-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
Keywords: ECMO; Cardiac arrest; Cardiopulmonary resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Out-of-hospital cardiac arrest on ECMO: Patients with out-of-hospital cardiac arrest indicated for ECMO
  Interventions: Procedure: Extracorporeal membrane oxygenation (ECMO)

INTERVENTIONS:
Procedure: Extracorporeal membrane oxygenation (ECMO) — In extracorporeal membrane oxygenation (ECMO), blood is pumped outside of the body to a heart-lung machine. The machine removes carbon dioxide and sends oxygen-rich blood back to the body. Blood flows from the right side of the heart to the heart-lung machine. It's then rewarmed and sent back to the body.

SUMMARY:
Cardiopulmonary resuscitation (CPR) for out-of-hospital cardiac arrest (OHCA) in specific cases could be improved by Extracorporeal membrane oxygenation (ECMO; ECPR). ECPR could be introduced in hospital after retrieval of an OHCA patient and also faster by implantation on scene. The aim is to verify the effectiveness of ECPR on scene in the Moravian-Silesian region.

DETAILED DESCRIPTION:
Patients undergoing cardiopulmonary resuscitation (CPR) for out-of-hospital cardiac arrest (OHCA) have a poor prognosis and a good long-term neurological outcome is achieved in about 10% of them. Extracorporeal membrane oxygenation (ECMO) can lead to an improvement in neurological outcome of up to 30% in a selected group of these critically ill patients. CPR for OHCA using ECMO in the hospital after patient admission (ECPR) is very demanding and depends on the best collaboration of pre-hospital care components with the hospital management. As good as the coordination of the different phases of care and transport is, patients often arrive to the hospital relatively late (over 60 minutes), and although the process of diagnosis and indication and ECMO implantation itself is rapid (approximately 15 minutes), the overall time from collapse to ECMO initiation is relatively long (over 60 minutes). It is this time, i.e. the duration of low organ perfusion during CPR, that may be the key parameter in determining the overall neurological outcome of treatment and prognosis of patients. Shortening this interval by having the ECMO team go to well-defined OHCA cases simultaneously with the ambulance car of the Emergency Department and connecting the patient to ECMO already in the field may lead to an improvement in the neurological outcome of the treatment of OHCA patients. In many locations abroad, this model is already used, and patients are connected to ECMO already in the field. Whether the model of field ECPR can be used in the Moravian-Silesian Region depends on a number of variables. These include the logic of information acquisition and selection of suitable patients, the logic of transporting the team and material to the scene, and the logic of connection with the provision of a safe and suitable environment for the ECMO implantation itself. The goal of this study is to validate the feasibility of the method on a simulated ECPR OHCA and further implant the mobile ECPR project in the Moravian-Silesian region.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Observed collapse and presumption of cardiac cause of cardiac arrest
* Estimated age up to 70 years
* Baseline rhythm of ventricular fibrillation or pulseless electrical activity (PEA)
* Basic bystander cardiopulmonary resuscitation (CPR), "bystander CPR", telephone assisted CPR (TANR)

Exclusion Criteria:

* Children or adults with estimated weight below 40 kg
* Known major comorbidities of the patient suggesting low rehabilitation potential (e.g. chronic obstructive pulmonary disease (COPD) IV, malignancy in tertiary phase)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after out-of-hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from cardiac arrest (collapse) to implantation of ECMO | up to 60 minutes
  The time from cardiac arrest (collapse) to implantation of ECMO will be recorded and assessed
Hospital mortality | up to 3 weeks
  Hospital mortality will be assessed for the period of 3 weeks
Cerebral Performance Category (CPC) score | 30 days
  Cerebral Performance Category (CPC) score will be observed 30 days after cardiac arrest
Neurological outcome (CPC score) | 6 months
  Neurological outcome will be assessed using the Cerebral Performance Category Scale (CPC) 6 months after cardiac arrest.
Neurological outcome (SF-36) | 6 months
  Neurological outcome will be assessed using the Short Form 36 Health Subject Questionnaire (SF-36) 6 months after cardiac arrest.
Neurological outcome (EQ-5D) | 6 months
  Neurological outcome will be assessed using the European Quality of Life Questionnaire (EQ-5D) 6 months after cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Burša, MD, PhD, EDEC, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - Emergency Medical Services, Moravian-Silesian Region, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.